CLINICAL TRIAL: NCT04676971
Title: Efficacy and Safety of Intravenously Administered hzVSF-v13 in Patients With COVID-19 Pneumonia: a Phase II, Proof of Concept, Multicentre, Randomized, Parallel-group, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of hzVSF-v13 in Patients With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmuneMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hzVSF_v13-0006
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100 mg hzVSF-v13 IV + SOC (Experimental): 100 mg hzVSF-v13 IV + SOC
  Interventions: Drug: hzVSF-v13
- 200 mg hzVSF-v13 IV + SOC (Experimental): 200 mg hzVSF-v13 IV + SOC
  Interventions: Drug: hzVSF-v13
- Placebo (saline) IV + SOC (Placebo Comparator): Placebo (saline) IV + SOC
  Interventions: Drug: Placebo (Normal saline solution)

INTERVENTIONS:
Drug: hzVSF-v13 — Dosage form: 100mg / 200mg of hzVSF-v13 (40 mg/mL in a 5 mL vial) Frequency: Dose at Day 1, 3, 7, D14(if necessary)
  Other Names: a humanized monoclonal antibody (mAb)
  Arms: 100 mg hzVSF-v13 IV + SOC; 200 mg hzVSF-v13 IV + SOC
Drug: Placebo (Normal saline solution) — Dosage form: 0.9% NaCl Solution Frequency: Dose at Day 1, 3, 7, D14(if necessary)
  Other Names: 0.9% Normal saline
  Arms: Placebo (saline) IV + SOC

SUMMARY:
Preliminarily investigate the safety and efficacy of two doses of hzVSF-v13 + SOC vs. placebo + SOC for the treatment of COVID-19 pneumonia.

DETAILED DESCRIPTION:
Proof of concept, multicentre, randomized, parallel-group, double-blind, placebo-controlled

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent from any patient capable of giving consent, or, when the patient is incapable of doing so, by his or her legal/authorized representative. Note: In accordance with the European Medicines Agency (EMA) "Guidance on the management of clinical trials during the covid-19 (coronavirus) pandemic version 3 28/04/2020", if written consent by the trial participant is not possible (for example because of physical isolation due to COVID-19 infection), consent may be given orally by the trial participant in the presence of an impartial witness.
2. Age 18 years or older.
3. Patient is currently hospitalized.
4. Diagnosis of COVID-19 pneumonia including a positive RT-PCR test for SARS-CoV-2 of any specimen and lung involvement confirmed with chest imaging (X-ray or computed tomography [CT] scan).
5. Able to comply with the study protocol.
6. Female patients must be postmenopausal (24 months of amenorrhea), surgically sterile or must agree to use an effective method of contraception throughout the study and for up to 120 days after stopping treatment. Effective contraception includes an established hormonal therapy or intrauterine device for females, and the use of a barrier contraceptive (i.e. diaphragm or condoms) with spermicide.

Exclusion Criteria:

1. Patients with known or suspected hypersensitivity to hzVSF-v13 or to any of its excipients.
2. Active tuberculosis or suspected active bacterial, fungal, viral, or other infection (besides COVID-19).
3. Anti-rejection or immunomodulatory drugs within the past 3 months.
4. Absolute neutrophil count (ANC) < 1000/µL at screening.
5. Platelet count < 50,000/ µL at screening.
6. ALT or AST > 5 x upper limit of normal (ULN) within 24 hours at screening.
7. Serum creatinine > 2 mg/dL (> 176.8 μmol/L) or estimated creatinine clearance < 30 ml/min measured or calculated by Cockroft Gault equation.
8. Pregnancy or breastfeeding.
9. Treatment with an investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization (approved/investigational COVID-19 antivirals and other off-label drugs recommended by local health authorities are permitted).
10. Patients who in the opinion of the treating physician should not participate in this program (ex: severe acute respiratory distress syndrome [ARDS], septicaemia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Clinical failure at Day 28 | Day 28
  A patient will be considered a clinical failure if on Day 28 the patient is dead, intubated and/or in ICU.

SECONDARY OUTCOMES:
Clinical Improvement, defined as a decrease of at least 2 points on the World Health Organization (WHO) ordinal scale | Day 28
  Clinical improvement is defined as a decrease of at least two points on the WHO ordinal scale from the Day 1 visit to the Day 28 visit.
Rate of overall survival (OS) at Day 28 and Day 60 | Day 28, Day 60
  Overall survival (OS), defined as the time from randomization to the date of death due to any cause, will be analysed by means of Kaplan-Meier methodology.
Incidence and severity of adverse events according to NCI CTCAE v5.0 | Day 60
  The incidence of AEs will be tabulated by MedDRA System Organ Class and Preferred Term. The incidence of AEs will also be summarised by System Organ Class, Preferred Term, and severity (based on NCI CTCAE v5.0 grades)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Sonnino, phD, Study Chair — OPIS s.r.l
Locations (9):
- Italy (2):
  - UOC Pneumologia, Bergamo
  - Dipartimento di Medicina Interna, Milan
- Russia (7):
  - Federal Siberian Scientific and Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk
  - Central City Hospital of Novoshakhtinsk, Novoshakhtinsk
  - SPb SBIH "Municipal Hospital №40", Saint Petersburg
  - Pokrovskaya Municipal Hospita, Saint Petersburg
  - Regional Clinical Hospital, Saratov
  - Regional Clinical Hospital No1, Smolensk
  - Federal State Budgetary Educational Institution of Higher Education, Ufa

IPD SHARING:
Plan to Share IPD: No